CLINICAL TRIAL: NCT06195553
Title: Application and Analysis of the Effectiveness of the STEPPS Program in Patients with BPD, Extending to Their Families with the Family Connections Program: a Randomized Controlled Trial
Brief Title: Application and Effectiveness of the STEPPS in Patients with BPD, Extending to Their Families with the FC Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Hospital de la Ribera (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STEPPSFCHULR
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: Personality disorder; borderline personality disorder; stepps; family connections; family focused therapy; family involvement; randomized controlled trial
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with one treatment condition and one control condition.
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEPPS for patients plus Family Connections for their families (Experimental): Intervention group that receives STEPPS program for patients to carry out the intervention about BPD symptoms and in parallel another group that receives Family Connectios program for their families to carry out the intervention about associated symptoms.
  Interventions: Behavioral: STEPPS plus Family Connections
- STEPPS for patients only (Active Comparator): Intervention group that receives STEPPS program for patients only to carry out the intervention about BPD symptoms.
  Interventions: Behavioral: STEPPS

INTERVENTIONS:
Behavioral: STEPPS plus Family Connections — The intervention will be based on cognitive and behavior treatment using STEPPS for the patients and dialectical and behavior treatment using Family Connections for the families. Main components STEPPS: psychoeducation, emotional regulation skills and behavioral regulation skills. Main components Family Connections: psychoeducation, skills training and peer support.
  Arms: STEPPS for patients plus Family Connections for their families
Behavioral: STEPPS — The intervention will be based on cognitive and behavior treatment using STEPPS for the patients. Main components STEPPS: psychoeducation, emotional regulation skills and behavioral regulation skills. Waiting list group: Participant's relatives of this group will be able to receive the Family Connections intervention after the research end.
  Arms: STEPPS for patients only

SUMMARY:
The present research project is framed within the issue of Borderline Personality Disorder (BPD). This condition stands as one of the most common challenges encountered within the mental health services of the National Health System. The primary objectives of this research are to verify whether the combined use of established treatments for patients and their families, conducted in parallel, leads to a greater improvement in patients and their families, respectively. Additionally, another aim of the project is to assess efficiency, defined as the acceptance of intervention programs by patients, their families, and clinical professionals, as well as to demonstrate their feasibility.

DETAILED DESCRIPTION:
The literature so far seems to indicate that involving family members in psychotherapeutic interventions for patients diagnosed with Severe Mental Disorders (SMD) such as psychosis or bipolar disorder is effective, reducing hospitalizations and increasing treatment satisfaction. However, interventions with such characteristics have not been found for patients with Borderline Personality Disorder (BPD), one of the disorders included under the umbrella of SMD. Therefore, it seems necessary to develop and implement comprehensive programs involving families, given the benefits observed in other SMD diagnoses such as psychosis or bipolar disorder.

BPD is one of the personality disorders that receives significant clinical attention and research, with suicide being one of the most associated problems with this diagnosis, ranging from 3-10%. The prevalence of BPD in the general population is considered to be around 1%, rising to 12% in clinical populations and 22% in hospitalized patients. Meta-analysis studies place Linehan's Dialectical Behavior Therapy (DBT) and Bateman and Fonagy's Mentalization-Based Therapy as the two interventions with the highest level of recommendation. Another widely supported intervention is Blum's Systems Training for Emotional Predictability and Problem Solving (STEPPS) program, especially effective when delivered in a group format within clinical and hospital settings due to its high adaptability. However, the issues described concerning patients with BPD inevitably lead to severe consequences in their work, emotional, and social environments. Relatives of individuals with BPD are more likely to experience psychological problems, burden, and depression. Generally, when family members participate in treatments, the patient's relapses decrease, recovery becomes easier, and overall family well-being improves. Presently, interventions for relatives of patients with BPD exist. Family Connections (FC) has received the most empirical support. Nevertheless, to date, there have been no studies analyzing whether adding intervention programs for family members contributes to an improvement in the STEPPS program, which is precisely the aim of this current research. Specifically, the objective of this work is to compare the effectiveness of the STEPPS protocol for patients with BPD and their relatives, compared to the STEPPS protocol for patients alone and the Family Connections program for their relatives.

The Randomized Clinical Trial (RCT) will be conducted following the guidelines of the Consolidated Standards of Reporting Trials (CONSORT: http://www.consort-statement.org) and the SPIRIT guidelines (Standard Protocol Items: Recommendations for Intervention Trials). Participants (N=120) will be randomly assigned to two groups (after receiving a diagnosis of Borderline Personality Disorder according to the DSM-5): 1) STEPPS program for patients 2) STEPPS program for patients and Family Connections for their relatives. Participants in the second group may receive the Family Connections intervention for their relatives after completing the research evaluation period for ethical reasons. Outcome measures will be assessed at baseline, post-treatment, and at 6-month follow-ups. About stadistical analysis, separate statistical analyses will be performed for caregivers and patients. Intent to treat analyses will be performed using Linear Mixed Models (LMMs). The clinical significance of change observed in the scores of outcome measures from one assessment moment (baseline) to another (post-treatment) will be determined calculating the Reliable Change Indexes.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Being at least 18 years old.
* Be a patients with symptoms compatible with a diagnosis of BPD who is undergoing treatment or follow-up in someone of the indicated recruitment centers.
* Sign an informed consent.

Exclusion Criteria:

* The presence of any pathology that prevents carrying out the intervention: major depression, psychosis, schizophrenia, substance dependence, eating disorders, another personality disorder, borderline IQ, etc., which due to its severity is currently interfering.

FAMILIES:

Inclusion Criteria:

* Being at least 18 years old.
* Be a relative of someone of the patients with symptoms compatible with a diagnosis of BPD who is undergoing treatment or follow-up in someone of the indicated recruitment centers.
* Sign an informed consent.

Exclusion Criteria:

* The presence of any pathology that prevents carrying out the intervention: major depression, psychosis, schizophrenia, substance dependence, eating disorders, another personality disorder, borderline IQ, etc., which due to its severity is currently interfering.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
BDI: Beck Depression Inventory (BDI-II; Beck, Steer, & Brown, 1996). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months
  This questionnaire assesses the degree of depressive symptomatology in the last week. It consists of 21 items rated on a scale from 0 (nothing) to 3 (very much).
OASIS: Overall Anxiety Severity and Impairment Scale (OASIS; Norman, Cissell, Means-Christensen, & Stein, 2006). Adapted into Spanish by Osma et al. (2019). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months
  This questionnaire assesses the degree of anxiety symptomatology in the last week. It consists of 5 items rated on a scale from 0 (mild) to 4 (extreme).
INQ: The Interpersonal Needs Questionnaire (INQ; Van Order et al., 2012). We will use the Spanish version by Marco & Pérez (2016). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the degree of interpersonal needs currently. It consists of 15 items rated on a scale from 1 (nothing true) to 7 (totally true).
ACWRSS: The Acquired Capability with Rehearsal for Suicide Scale (ACWRSS; George et al., 2016). We will use the Spanish version by Marco et al. (2020). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the acquired capability with rehearsal for suicide. It consists of 7 items rated on a scale from 0 (disagreement) to 8 (agreement).
DERS: Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2008). We will use the Spanish version by Hervás & Jódar (2008). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the ability to regulate emotions. It consists of 28 items rated on a scale from 1 (hardly never) to 5 (almost always).
BSL-23: Borderline Symptom List 23 (BSL-23; Bohus et al., 2008). We will use the Spanish version by Feliú-Soler et al. (2012). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the degree of symptoms of borderline personality disorders in the last week. It consists of 23 items rated on a scale from 0 (never) to 4 (very much) and 11 items rated on a scale from 0 (nothing) to 4 (daily).
QLI: Quality of Life Index (QLI; Ferrans & Powers, 1985). We will use the Spanish version by Mezzich et al. (2000). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the level of quality of life currently. It consists of 10 items rated on a scale from 1 (bad) to 10 (excellent).
PIL-20: Purpose in Life-20 (PIL-20; Crumbaugh & Maholick, 1964). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the purpose in life. It consists of 20 items rated on a scale from 1 (nothing) to 7 (very much).
VIRS: Validating and Invalidating Responses Scale (VIRS; Fruzzetti, 2007). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the degree of validated or invalidating responses from the family in the last week. It consists of 15 items rated on a scale from 0 (never) to 4 (almost every time).
LEAP: Lum Emotional Availability of Parents (LEAP; Lum & Phares, 2005). | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the perception of emotional availability from the parents. It consists of 15 items rated on a scale from 0 to 6 about the father and 0 to 6 about the mother.
Registry of family-patient critical incidents in the last three months. | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  The registry consist of 6 questions about number of critical incidents such as suicide attempts or visits to the emergency room.

SECONDARY OUTCOMES:
BAS: Burden Assessment Scale (BAS; Reinhard et al., 1994). Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the level of disease burden in the last 6 months. It consists of 19 items rated on a scale from 1 (nothing) to 4 (very much).
FES: Family Empowerment Scale (FES; Koren, DeChillo, & Friesen, 1992). Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the degree of perception of mastery and empowerment. It consists of 34 items rated on a scale from 1 (totally false) to 4 (totally true).
DASS-21: Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995). We will use the Spanish version by Bados, Solanas, & Andrés (2005). Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the degree of depression, anxiety and stress in the last week. It consists of 21 items rated on a scale from 0 (never) to 3 (very much).
QLI: Quality of Life Index (QLI; Ferrans & Powers, 1985). We will use the Spanish version by Mezzich et al. (2000). Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the level of quality of life currently. It consists of 10 items rated on a scale from 1 (bad) to 10 (excellent).
SVSI-Q: The Self-Validation and Self-Invalidation Questionnaire (SVSI-Q; Fruzzetti & Davis, in preparation). Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the degree of self-validation or self-invalidation. It consists of 24 items rated on a scale from 1 (hardly ever) to 5 (always).
PIL-20: Purpose in Life-20 (PIL-20; Crumbaugh & Maholick, 1964). Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the purpose in life. It consists of 20 items rated on a scale from 1 (nothing) to 7 (very much).
Measurement of acceptance and satisfaction. Treatment Opinion Scale (adapted from Borkovec & Nave, 1972). Relatives's responses | immediately after treatment, also at follow-up assessment periods (6 months)
  This questionnaire assesses the opinión about treatment at the end of the investigation. It consists of 7 items rated on a scale from 1 (nothing) to 7 (very much).
Registry of family-patient critical incidents in the last three months. Relatives's responses | At the beginning of the intervention and immediately after treatment, also at follow-up assessment periods (6 months)
  The registry consist of 6 questions about number of critical incidents such as suicide attempts or visits to the emergency room.

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, Psychology, Study Director — Universidad Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajalin M, Wickholm-Pethrus L, Hursti T, Jokinen J. Dialectical behavior therapy-based skills training for family members of suicide attempters. Arch Suicide Res. 2009;13(3):257-63. doi: 10.1080/13811110903044401. PMID 19590999
- [Background] Liljedahl SI, Kleindienst N, Wangby-Lundh M, Lundh LG, Daukantaite D, Fruzzetti AE, Westling S. Family Connections in different settings and intensities for underserved and geographically isolated families: a non-randomised comparison study. Borderline Personal Disord Emot Dysregul. 2019 Aug 26;6:14. doi: 10.1186/s40479-019-0111-6. eCollection 2019. PMID 31463066
- [Background] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Background] Flynn D, Kells M, Joyce M, Corcoran P, Herley S, Suarez C, Cotter P, Hurley J, Weihrauch M, Groeger J. Family Connections versus optimised treatment-as-usual for family members of individuals with borderline personality disorder: non-randomised controlled study. Borderline Personal Disord Emot Dysregul. 2017 Aug 30;4:18. doi: 10.1186/s40479-017-0069-1. eCollection 2017. PMID 28861273
- [Background] Fernandez-Felipe I, Guillen V, Marco H, Diaz-Garcia A, Botella C, Jorquera M, Banos R, Garcia-Palacios A. Efficacy of "Family Connections", a program for relatives of people with borderline personality disorder, in the Spanish population: study protocol for a randomized controlled trial. BMC Psychiatry. 2020 Jun 15;20(1):302. doi: 10.1186/s12888-020-02708-8. PMID 32539740
- [Background] Dixon L, McFarlane WR, Lefley H, Lucksted A, Cohen M, Falloon I, Mueser K, Miklowitz D, Solomon P, Sondheimer D. Evidence-based practices for services to families of people with psychiatric disabilities. Psychiatr Serv. 2001 Jul;52(7):903-10. doi: 10.1176/appi.ps.52.7.903. PMID 11433107
- [Background] undefined